CLINICAL TRIAL: NCT05765981
Title: An Open, Dose-escalating Early Clinical Trial to Evaluate the Tolerability, Safety, and Efficacy of VGN-R09b by Intra Striatum Injection in Patients With Aromatic L-amino Acid Decarboxylase (AADC) Deficiency.
Brief Title: An Early Clinical Trial to Evaluate VGN-R09b for Treatment of Aromatic L-amino Acid Decarboxylase (AADC) Deficiency.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Vitalgen BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGN-R09b-001
Record Dates: First submitted 2023-01-18; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Aromatic L-amino Acid Decarboxylase (AADC) Deficiency
Keywords: AADC, AAV9, CNS gene therapy
MeSH Terms: conditions — Aromatic amino acid decarboxylase deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aromatic L-amino acid decarboxylase (AADC) deficiency (Experimental): This early Phase trial is to prove the safety and efficacy of VGN-R09b to treat patients with AADC deficiency.
  Interventions: Drug: VGN-R09b

INTERVENTIONS:
Drug: VGN-R09b — VGN-R09b will be injected into bilateral putamen by stereotactic surgery.（Through the SmartFlow Ventricular Cannula or the parenchymal injection tube actually used in the research center）

SUMMARY:
This early Phase trial is to prove the safety and efficacy of VGN-R09b to treat patients with AADC deficiency.

DETAILED DESCRIPTION:
Aromatic L-amino acid decarboxylase (AADC) is an enzyme responsible for the final step in the synthesis of neurotransmitters dopamine and serotonin. AADC deficiency is a rare genetic disorder. VGN-R09b is a kind of Gene therapy with adeno-associated virus (AAV) serotype 9 (AAV9) driven human AADC (hAADC) being injected directly into striatum.

This is a single-center, open, dose-climbing investigator-sponsored early-stage clinical study that included a dose-climbing phase and a dose-expanding phase.

This study is to give preliminary evidence for the safety and efficacy of VGN-R09b treatment for patients with Aromatic L-amino acid decarboxylase (AADC) deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. The child patient has to be ≥2 years old and < 8 years old, or a head circumference big enough for surgery.
2. Historical diagnosis of AADC deficiency with clinical symptoms consistency, AND confirmed by one of the lab tests: (1) CSF neurotransmitter profile demonstrating reduced HVA and 5-HIAA, and elevated L-Dopa concentrations; (2) Plasma AADC activity less than or equal to 5 pmol/min/mL, AND with Molecular genetic confirmation of homozygous or compound heterozygous mutation of IVS6+4A>T in DDC.
3. Motor development at baseline ≤3 months, and Failed to benefit from standard medical therapy (dopamine agonists, monoamine oxidase inhibitor or related form of Vitamin B6) at discretion of investigators.
4. Stable medication regimen for treatment of AADC deficiency: (i.e. no new medications introduced for at least 6 months, and no existing medication dose changes for at least 3 months prior to Baseline).
5. Parent(s)/legal guardian(s) with custody of subject must give their consent for subject to enroll in the study
6. Parent(s)/legal guardian(s) of the subject must agree to comply with the requirements of the study, including providing disease information and support disease assessment of symptoms.

Exclusion Criteria:

1. Intracranial neoplasm or any structural brain abnormality or lesion (e.g., severe brain atrophy, white matter degenerative changes), which, in the opinion of the study investigators, would confer excessive risk and/or inadequate potential for benefit.
2. Presence of other significant medical or neurological conditions that would create an unacceptable operative or anesthetic risk (including congenital heart disease, respiratory disease with home oxygen requirement, history of serious anesthesia complications during previous elective procedures, history of cardiorespiratory arrest), liver or renal failure, malignancy, or HIV positive.
3. Severe coagulopathy, or need for ongoing anticoagulant therapy.
4. clinically active infection or with severe infection within 12 weeks before screening (e.g. adenovirus or herpes virus, pneumonia, sepsis, central nervous system infection).
5. Previous stereotactic neurosurgery, or any gene/cell therapy.
6. Received live vaccination within 4 weeks.
7. Patients with anti-AAV9 neutralizing antibody titer over 1,200 folds.
8. Contraindication to sedation during surgery or imaging studies (PET or MRI).

Ages: 24 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2029-02-20 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs), Serious Adverse Events (SAEs) | Week 52
  Number of Adverse Events (AEs), Serious Adverse Events (SAEs)
Achievement Ratio of the four motor development milestones (Head control, Sit independently, Stand/stepping with support and Walk with minimal assistant) | Week 52
  Achievement Ratio of the four motor development milestones (Head control, Sit independently, Stand/stepping with support and Walk with minimal assistant) according to PDMS-II score.

CONTACTS AND LOCATIONS:
Overall Officials: Jiwen Wang, Doctor, Study Chair — Shanghai Children's Medical Center, affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Children's Medical Center Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, No. 1678, Dongfang Road, Pudong New Area, Shanghai, China